CLINICAL TRIAL: NCT06727084
Title: Predictive Value of Serum Albumin in Patients With Acute Coronary Syndrome
Brief Title: Serum Albumin in Acute Coronary Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Magdy Adel Zaki, Internal medicine Resident, Sohag University
Other Study IDs: Soh-Med--24-11-04MS
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Serum Albumin in Patients With Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aims to investigate the predictive value of serum albumin and short-term mortality in patients with Acute Coronary Syndrome (ACS)

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) refers to a group of conditions that include ST-elevation myocardial infarction (STEMI), non-ST elevation myocardial infarction (NSTEMI), and unstable angina. It is a type of coronary heart disease (CHD), which is responsible for one-third of total deaths in people older than 35. Some forms of CHD can be asymptomatic, but ACS is always symptomatic .

Long-term mortality remains high in patients presenting with ACS despite advances in diagnosis and treatment. Therefore, identification of high-risk patients in this patient group is of prime importance. To date, various risk scores and biomarkers have been used for this purpose .

Albumin is the major protein in human plasma and the most abundant protein in the extracellular compartment. Albumin has multiple important physiological functions including maintenance of plasma osmotic pressure and capillary permeability, a ligand for many endogenous and exogenous compounds and it also affects the pharmacokinetics of several drugs .

In addition, low serum albumin is associated with increased adverse clinical outcomes and prognosis in cancer, heart failure, stroke, and stable coronary artery disease (CAD). Similarly, in patients with ACS, presence of hypoalbuminemia has been associated with increased severity of coronary lesions, no-reflow, increased in-hospital, and long-term mortality as well as development of heart failure .

Until now, several studies have documented the prognostic value of SA in patients with stable coronary artery disease (CAD), ST elevation myocardial infarction, and pulmonary embolism. In this research, the authors also concluded that admission SA level was a strong and independent predictor of all-cause long-term mortality in patients with ACS. Although the research was interesting and well-conducted, we have some comments .

Current European and North American guidelines recommend risk stratification of ACS cases using available risk scores, such as the thrombolysis in myocardial infarction (TIMI) score and the Global Registry of Acute Coronary Events (GRACE) score, to determine the in-hospital and 6-months risk of death and myocardial infarction in patients with ACS following an index event

. Beside that, a recent study revealed that these scores had an adequate predictive power for long-term mortality in patients who were diagnosed and hospitalized with ACS .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who were admitted to the emergency department or coronary care unit with a diagnosis of acute coronary syndrome (ACS) will be eligible for inclusion.

Exclusion Criteria:

1. Patients with a history of chronic liver disease, nephrotic syndrome, or other conditions known to affect serum albumin levels.
2. Patients receiving albumin infusions or other treatments that could potentially interfere with serum albumin levels.
3. Patients with incomplete medical records or missing laboratory data.
4. Patients who declined to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who were admitted to the emergency department or coronary care unit with a diagnosis of acute coronary syndrome (ACS) will be eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Value of Serum Albumin in Patients With Acute Coronary Syndrome | 12 week after the end of treatment
  low serum albumin is associated with increased adverse clinical outcomes and prognosis in cancer, heart failure, stroke, and stable coronary artery disease (CAD). Similarly, in patients with ACS, presence of hypoalbuminemia has been associated with increased severity of coronary lesions, no-reflow, increased in-hospital, and long-term mortality as well as development of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Osama A Arafa, Professor, Study Director — Faculty of Medicine Sohag University; Hamdy S Mohamed, A .Professor, Study Director — Faculty of Medicine Sohag University; Ahmed E Ebrahim, Lecturer, Study Director — Faculty of Medicine Sohag University
Locations (1):
- Faculty of medicine Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien SC, Chen CY, Leu HB, Su CH, Yin WH, Tseng WK, Wu YW, Lin TH, Chang KC, Wang JH, Wu CC, Yeh HI, Chen JW. Association of low serum albumin concentration and adverse cardiovascular events in stable coronary heart disease. Int J Cardiol. 2017 Aug 15;241:1-5. doi: 10.1016/j.ijcard.2017.04.003. Epub 2017 Apr 7. PMID 28413113
- [Background] Polat N, Oylumlu M, Isik MA, Arslan B, Ozbek M, Demir M, Kaya H, Toprak N. Prognostic Significance of Serum Albumin in Patients With Acute Coronary Syndrome. Angiology. 2020 Nov;71(10):903-908. doi: 10.1177/0003319720941747. Epub 2020 Jul 17. PMID 32677445
- [Background] D'Ascenzo F, Biondi-Zoccai G, Moretti C, Bollati M, Omede P, Sciuto F, Presutti DG, Modena MG, Gasparini M, Reed MJ, Sheiban I, Gaita F. TIMI, GRACE and alternative risk scores in Acute Coronary Syndromes: a meta-analysis of 40 derivation studies on 216,552 patients and of 42 validation studies on 31,625 patients. Contemp Clin Trials. 2012 May;33(3):507-14. doi: 10.1016/j.cct.2012.01.001. Epub 2012 Jan 11. PMID 22265976
- [Background] Zegre-Hemsey JK, Asafu-Adjei J, Fernandez A, Brice J. Characteristics of Prehospital Electrocardiogram Use in North Carolina Using a Novel Linkage of Emergency Medical Services and Emergency Department Data. Prehosp Emerg Care. 2019 Nov-Dec;23(6):772-779. doi: 10.1080/10903127.2019.1597230. Epub 2019 Apr 17. PMID 30885071